CLINICAL TRIAL: NCT00744809
Title: A Phase I, Double-blind, Double-dummy, Randomized, Placebo Controlled and Active Controlled Trial to Evaluate the Effect of TMC278 25 mg Daily at Steady-state and the Effect of Efavirenz (EFV) 600 mg Daily at Steady-state on the QT/QTc Interval, in 2 Randomized Panels of Healthy Volunteers
Brief Title: TMC278-TiDP6-C152: A Study to Assess the Effects of TMC278 and Efavirenz (EFV) on the QT/QTc Interval (Heart Conduction and Heart Rhythm) in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CR015088
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-03

CONDITIONS: Human Volunteers
Keywords: TMC278-C152; TMC278-TiDP6-C152; Healthy Volunteers; QT/QTc interval
MeSH Terms: interventions — Rilpivirine; Moxifloxacin; efavirenz

INTERVENTIONS:
Drug: TMC278; Moxifloxacin; Efavirenz

SUMMARY:
This is a study to evaluate the effect of TMC278 25 mg daily on the QT/QTc interval (heart conduction and heart rhythm) in healthy volunteers. In a separate panel of healthy volunteers, the effect of efavirenz (EFV) 600 mg daily on the QT/QTc interval will be evaluated.

DETAILED DESCRIPTION:
This is a trial to evaluate the effect of TMC278 25 mg daily on the QT/QTc interval (heart conduction and heart rhythm) in healthy volunteers. In a separate panel of healthy volunteers, the effect of efavirenz (EFV) 600 mg daily on the QT/QTc interval will be evaluated. TMC278 is being investigated as a treatment for HIV-1 infection. In one panel, the effect of TMC278 at steady-state on the QT/QTc interval in healthy volunteers will be evaluated in a double-blind (neither the doctor nor the patient know if the patient is getting active drug or placebo), randomized (study drug assigned by chance), placebo controlled and positive controlled 3-way crossover design. One dose regimen of 25 mg daily of TMC278 will be tested for 11 days. In a second session, a single dose of 400 mg of moxifloxacin will be used as a positive control to assess trial sensitivity. A placebo session will be included as a reference. In a separate panel, the effect of EFV at steady-state on the QT/QTc interval in healthy volunteers will be evaluated in a double-blind, randomized, placebo controlled 2-way crossover design. One dose regimen of 600 mg daily of EFV will be tested for 11 days. Similar to the TMC278 panel, a placebo session will be included as a reference. The overall trial population will consist of 120 healthy volunteers of which at least 30% and no more than 50% are female and of which at least 20% are non-Hispanic Caucasians. Patients will be randomized in a 1:1 ratio to either the TMC278 panel or the EFV panel. The randomization between the 2 panels will be stratified by gender and ethnicity and the randomization within each panel will be stratified by gender. Each patient in the TMC278 panel will receive in 3 sessions in a random order: TMC278 25 mg daily on Day 1-11 and moxifloxacin placebo q.d. on Day 11 (Treatment A), TMC278 placebo daily on Day 1-11 and moxifloxacin placebo q.d. on Day 11 (Treatment B), and TMC278 placebo daily on Day 1-11 and moxifloxacin 400 mg q.d. on Day 11 (Treatment C). All intakes of TMC278, moxifloxacin, TMC278 placebo and moxifloxacin placebo will be under fed conditions and will take place under supervision in the unit. There will be a washout period of at least 21 days between consecutive treatments. Each patient in the EFV panel will receive in 2 sessions in a random order: EFV 600 mg daily for 11 days (Treatment D) or EFV placebo q.d. for 11 days (Treatment E). All intakes of EFV and EFV placebo will be under fasted conditions and will take place under supervision in the unit. There will be a washout period of at least 53 days between the 2 treatments. In both the TMC278 and the EFV panels, ECGs will be recorded continuously for 24 hours by Holter monitoring on Day -1 and Day 11 of all treatment sessions. In addition, for safety monitoring, 12-lead ECGs will be performed at predefined time points. Pharmacokinetic samples will be collected on Day -1, Day 9, Day 10, and Day 11, within 5 minutes after safety ECG recording or Holter extraction time point, if applicable, for the determination of TMC278, moxifloxacin or EFV plasma concentrations, as appropriate. Safety and tolerability will be monitored throughout the trial. In the TMC278 Panel, TMC278 or placebo will be given by mouth on Days 1-11 and Moxifloxican or placebo will be given by mouth on Day 11. Patients will return after each washout period for a total of 3 cycles. In the EFV Panel, EFV or placebo will be given by mouth on Days 1-11. Patients will return after the washout period for a total of 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must: be non-smokers (no tobacco products, nicotine or nicotine containing products of any kind for at least 1 year)
* have a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* be healthy on the basis of a pre-trial physical examination, medical history, electrocardiogram, vital signs and the results of routine blood and urine tests at screening
* have a normal 12-lead ECG at screening and on Day -1 (safety ECG) of the first treatment period.

Exclusion Criteria:

* Patients must not: have a positive HIV-1 or -2 test at trial screening
* be a female of childbearing potential without the use of effective birth control methods or not willing to continue practicing these birth control methods from screening onwards until at least 30 days after last intake of trial medication
* have a history or evidence of current use of alcohol, barbiturate, amphetamine, recreational, or narcotic drug use
* have Hepatitis A, B or C infection at trial screening
* have participated in an investigational drug trial within 60 days prior to the first intake of trial medication
* have a history of clinically relevant heart rhythm disturbances
* have blood pressure (BP) outside of normal range (sitting systolic blood pressure <90 or >140 mmHg and/or diastolic blood pressure <40 or >90 mmHg) at screening or on Day -1 of the first treatment period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of TMC278 25 mg daily at steady state on the QT/QTc interval in healthy volunteers.

SECONDARY OUTCOMES:
To evaluate steady-state PK of TMC278 25 mg daily in healthy volunteers; to evaluate the effect of EFV 600 mg daily and separately, a single dose of moxifloxican (400 mg) at steady state, on the QT/QTc interval in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: Clinical Study Report Synopsis of TMC278-TiDP6-C152: A study to assess the effects of TMC278 and Efavirenz (EFV) on the QT/QTc interval (heart repolarization) in healthy volunteers. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1010&filename=CR015088_CSR.pdf